CLINICAL TRIAL: NCT03815539
Title: Correlation of Noninvasive Tear Film Function and the Optical Quality in Mild and Moderate Dry Eye
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jin Yuan (Other)
Responsible Party: Sponsor-Investigator, Jin Yuan, Professor, Zhongshan Ophthalmic Center, Sun Yat-sen University
Organization: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 20181230
Record Dates: First submitted 2018-01-15; First posted 2019-01-24 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2018-01

CONDITIONS: Tear Film Insufficiency; Dry Eye
Keywords: dry eye; noninvasive tear breakup time; tear film related optical quality; correlation analysis
MeSH Terms: conditions — Xerophthalmia; Dry Eye Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- dry eye group (Experimental): Part of the subjects will be instilled with one drop of 0.1% sodium hyaluronate in one of their eyes, then they will be tested with the devices of Oculus Keratograph 5M and Optical Quality Analysis SystemⅡ at different time points (10min, 30min, 60min, 90min and 120min).
  Interventions: Device: 0.1% sodium hyaluronate

INTERVENTIONS:
Device: 0.1% sodium hyaluronate — In dry eye group, part of the subjects will be instilled with one drop of 0.1% sodium hyaluronate in one of their eyes, then they will be tested with the devices of Oculus Keratograph 5M and Optical Quality Analysis SystemⅡ at different time points (10min, 30min, 60min, 90min and 120min).

SUMMARY:
2017 International Dry Eye Workshop (DEWS) defines dry eye as a multifactorial ocular surface disease characterized by tear film instability with disturbed visual function. As a smooth transparent structure and the outmost layer of the whole ocular refractive system, tear film plays an important role. In dry eye, the instability of tear film caused by a lack of tear volume or high evaporation makes it more vulnerable to break up during blinking intervals, exposing the rough epithelium of the corneal surface and introducing extra aberrations and scatter. This would affect image sharpness on the retina and lower the optical quality. Also, it had been observed that the dynamic tear film scattering was reduced and the objective optical quality was improved transiently after artificial tears instillation. Though these findings supported the fact of visual quality impairment in dry eye. It remains unclear how does the tear film instability affect the visual quality in specific. Whether it lowers the optical quality of the whole ocular or just affects the tear-film associated part alone and whether there is a correlation with the tear film function are still unknown and to be answered. So we wondered whether there is a correlation between the tear film function and the related optical quality in dry eye. Though it had been inspected that the invasive tear break up time by fluorescein staining was positively correlated with the related scattering of tear film. To the newest dry eye diagnosis criteria of 2017 DEWS, the non-invasive tear break-up time has been amended to the first line instead of the invasive methods, e.g. fluorescein staining, which was thought to be less accurate and less credible. What's more, the invasive method of tear film evaluation might introduce confounding factors to the successive optical quality assessment. So we need a more accurate investigation to the relationships of the tear film function and the optical quality in dry eye. This study was intended to measure the non-invasive tear break-up time and the objective optical quality in normal people and dry eye patients to illustrate this question. In addition, we will investigate the relation of evolution trends of NIKBUT and objective optical quality under artificial tears for a better illustration.

DETAILED DESCRIPTION:
According to the 2017 International Dry Eye Workshop (DEWS), dry eye is "a multifactorial disease of the ocular surface characterized by ocular symptoms, in which tear film instability and hyperosmolarity, ocular surface inflammation and damage, and neurosensory abnormalities play etiological roles." Among the various symptoms, blurred vision and vision fluctuation are quite common, especially after long time reading or screen work. While the vision discomfort might point to visual quality impairment in dry eye. As the most outlayer and smooth transparent structure of the ocular, tear film plays an important role in the whole ocular refraction. In dry eye patients, the instability of tear film caused by lack of tear volume or high evaporation makes it more vulnerable to break out during blinking intervals and expose the rough epithelium of the corneal surface, which would introduce extra aberration and scattering. While the extra scattering would affect the image sharpness projected to the retina and might lower down the optical quality. Moreover, the more distant the scattering source, the more effects on retina image and optical quality. Indeed, it had been proved that compared with normal people, the whole ocular scattering was higher and the optical quality was lower in dry eye. Also, it had been observed that the dynamic tear film scattering was reduced and the objective optical quality was improved transiently after artificial tears instillation. Though these findings supported the fact of visual quality impairment in dry eye. It remains unclear how does the tear film instability affect the visual quality in specific. Whether it lowers the optical quality of the whole ocular or just affects the tear-film associated part alone and whether there is a correlation with the tear film function are still unknown and to be answered. So we wondered whether there is a correlation between the tear film function and the related optical quality in dry eye. Though it had been inspected that the invasive tear break up time by fluorescein staining was positively correlated with the related scattering of tear film. To the newest dry eye diagnosis criteria of 2017 DEWS, the non-invasive tear break-up time has been amended to the first line instead of the invasive methods, e.g. fluorescein staining, which was thought to be less accurate and less credible. What's more, the invasive method of tear film evaluation might introduce confounding factors to the successive optical quality assessment. So we need a more accurate investigation to the relationships of the tear film function and the optical quality in dry eye. This study was intended to measure the non-invasive tear break-up time and the objective optical quality in normal people and dry eye patients to illustrate this question. In addition, we will investigate the relation of evolution trends of NIKBUT and objective optical quality under artificial tears for a better illustration.

ELIGIBILITY:
Inclusion Criteria:

* for dry eye group: Ocular Surface Disease Index (OSDI) between 13 to 32 and NIBUT <10 seconds.
* for normal group: in absence of ocular symptoms or signs.

Exclusion Criteria:

* opacity of the refractive tissue
* history of ocular surgery that might affect the tear film (eg, refractive surgery, punctum plug insertion, etc)
* best corrected visual acuity of decimal vision < 1.0
* spherical error ≥ 6 diopters (D)
* cylindrical error ≤-2.0 D or ≥+2.0D
* allergy to the 0.1% sodium hyaluronate
* any condition that might interfere with the optical quality.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-06-30 (Actual); Primary Completion 2019-12-28 (Estimated); Study Completion 2019-12-28 (Estimated)

PRIMARY OUTCOMES:
The difference of tear film function as NIBUT by Keratograph 5M between dry eye and normal group | One day visit
  Keratograph 5M was used for NIBUT to test in the dry eye and normal group for tear film function.
The difference of the optical quality as scattering index between dry eye and normal group | One day visit
  The scattering index by OQAS for optical quality was tested in dry eye and normal group.
The correlation of NIBUT and scattering index in normal group | One day visit
  Pearson correlation was tested between NIBUT and scattering index in normal group.
The correlation of NIBUT and scattering index in dry eye group | One day visit
  Pearson correlation was tested between NIBUT and scattering index in dry eye group.
Time changing pattern of NIBUT and scattering index in dry eye group | base line, 10, 30,60, 90, 120 min after 0.1% sodium hyaluronate instillation
  The NIBUT and the scattering index change was tested before and after 0.1% sodium hyaluronate instillation in dry eye group

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-Sen University, Guangzhou, Guangdong, China